CLINICAL TRIAL: NCT06750601
Title: Rehablines: a Further Use Databank to (re)Use Routine Clinical Data for Scientific Research in Rehabilitation of People With Physical Disabilities and/or Chronic Diseases
Acronym: Rehablines
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: UMCG RR number: 16881
Record Dates: First submitted 2024-12-09; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Within the Center of Rehabilitation multidisciplinary treatment is provided to people with various physical disabilities and/or chronic diseases. During and in the context of this treatment, a lot of data is routinely collected. Rehablines is initiated to re-use this routine clinical data in a database for future scientific research. Rehablines aims to: - Efficiently conduct high quality scientific research aimed at patient characteristics, underlying disease processes, and treatment effects; - Provide insight into (short and long-term) treatment effects and efficiency of these rehabilitation treatments; - Personalize treatment by comparing data from the individual patient with data from a large number of patients with similar characteristics from Rehablines.

ELIGIBILITY:
Inclusion Criteria:

* all participants receiving care at the Center for Rehabilitation of the University Medical Center Groningen

Exclusion Criteria:

* n.a.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In the UMCG-CvR rehabilitation care is provided to patients with a variety of physical disabilities and/or chronic diseases. Provided types of rehabilitation include for instance neurorehabilitation, orthopedic rehabilitation, oncology rehabilitation, pain rehabilitation, pediatric rehabilitation and rehabilitation in chronic illnesses, e.g. heart, lung, diabetes, thoracic and transplant rehabilitation. All patients who are starting their treatment in our facility are invited to participate in Rehablines.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2044-01 (Estimated); Study Completion 2044-01 (Estimated)

PRIMARY OUTCOMES:
Clinical data | Timepoint 1: pre-treatment. Timepoint 2: throughout study completion (on average 12 weeks). Timepoint 3: up to 1 year follow up
  Rehablines is a unique databank that purely re-uses clinical data for research. All data that is collected during the treatment of our patients can be re-used with patient consent.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Rehabilitation of the University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Kammen K, Krops LA, Geertzen JHB, Dekker R. Rehablines: a Dutch further use databank to (re)use routine real world clinical data for scientific research in rehabilitation of people with physical disabilities and/or chronic diseases - a cohort profile. BMJ Open. 2025 Aug 8;15(8):e099089. doi: 10.1136/bmjopen-2025-099089. PMID 40780713